CLINICAL TRIAL: NCT04409574
Title: COVID19 Viral Clearance Among the Infected Healthcare Workers In Assiut University Hospitals
Brief Title: COVID 19 Viral Clearance Among the Infected Healthcare Workers In Assiut University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Roshdy Elkhayat, lecturer, Assiut University
Other Study IDs: COVID19 among HCWs
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Infection, Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — * Complete Blood Count (CBC) by (Pentra 80 Horiba blood counter).
  * Erythrocyte Sedimentation Rate (ESR) by westergren method.
  * Liver function , Kidney function tests, triglyceride , LDH, CK, CK-MB Na, K, Mg, Phosphorus, Ca, CRP, Ferritin ) (Dimension RXLautomated blood chemistry analyser).
  * HCV Ab, HBsAg and HIV Ag-Ab on Abott Architect i1000R
  * Prothrombin time , concentration, INR and D-Dimerand on sysmex 1500 corona virus investigation: Viral RNA extraction by Qiagen viral RNA extraction large volume: on QiAcube extractor
    * Coronavirus (Covid -19) genesig Real time PCR assay : on 7500 fast Applied biosystem
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This work was aimed to determine the time of COVID 19 viral clearance in healthcare workers, assessment of clinical presentation and severity of COVID 19 infection among healthcare workers and discover relation between the time of COVID 19 viral clearance resolution of symptoms

DETAILED DESCRIPTION:
COVID-19 has been spreading rapidly globally, with a considerable impact on global morbidity, mortality and healthcare utilization. This viral disease is caused by the Coronaviruses (CoV) which belong to the genus'coronavirus' of the Coronaviridae family.

Coronaviruses are enveloped positive strand RNA viruses with the largest known RNA genomes-30-32 kb-with a 50 -cap structure and 30 -poly-A tail (Lei et al.2018). The transcription works through the replication-transcription complex (RCT) organized in double-membrane vesicles and via the synthesis of subgenomic RNAs (sgRNAs) sequences. Of note, transcription termination occurs at transcription regulatory sequences, located between the so-called open reading frames (ORFs). In the atypical CoV genome, at least six ORF scan could be present (Woo et al., 2020) .

Health workers are at the front line of the COVID-19 outbreak response and as such are exposed to hazards that put them at risk of infection (Li e al.,2020). thus keeping the implementation of infection prevention and control (IPC) and its knowledge and practice are of great importance in healthcare settings to protect them from infections (Wang et al., 2020).

ELIGIBILITY:
Inclusion Criteria:

* Covid 19 infected healthcare workers.

Exclusion Criteria:

* Risky healthcare workers (diabetic hypertensive and more than 50 years)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Covid 19 infected healthcare workers in Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
the time of Covid 19 viral clearance in medical healthcare workers and its relation to clinical presentation, severity among and resolution of symptoms. | basline
  different relations between different symptoms, investigation results and time of viral clearness

SECONDARY OUTCOMES:
knowledge and practice of infection control measures | baseline
  good and bad knowledge or practice

REFERENCES:
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] Lei J, Kusov Y, Hilgenfeld R. Nsp3 of coronaviruses: Structures and functions of a large multi-domain protein. Antiviral Res. 2018 Jan;149:58-74. doi: 10.1016/j.antiviral.2017.11.001. Epub 2017 Nov 8. PMID 29128390
- [Background] Wang J, Zhou M, Liu F. Reasons for healthcare workers becoming infected with novel coronavirus disease 2019 (COVID-19) in China. J Hosp Infect. 2020 May;105(1):100-101. doi: 10.1016/j.jhin.2020.03.002. Epub 2020 Mar 6. No abstract available. PMID 32147406
- [Background] Woo PCY, Huang Y, Lau SKP, Yuen KY. Coronavirus genomics and bioinformatics analysis. Viruses. 2010 Aug;2(8):1804-1820. doi: 10.3390/v2081803. Epub 2010 Aug 24. PMID 21994708